CLINICAL TRIAL: NCT06065501
Title: Frailty Trajectories and Effects of Personalized Actionable Connected Extensible (PACE) Interventions Among Patients With Chronic Kidney Disease: A Longitudinal Study
Brief Title: Effects of Personalized Actionable Connected Extensible (PACE) Interventions Among Patients With Chronic Kidney Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Cheng Kung University (Other)
Responsible Party: Principal Investigator, Miaofen Yen, Professor, Department of Nursing College of Medicine, National Cheng Kung University, National Cheng Kung University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: B-ER-109-494
Record Dates: First submitted 2023-09-26; First posted 2023-10-04 (Actual); Results first posted 2025-06-26 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: CKD - Chronic Kidney Disease
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PACE intervention (Experimental): The intervention group (PACE intervention) utilizes mobile social network support, employing a LINE group to implement a personalized plan based on the TTM model for establishing a care program.
  Interventions: Behavioral: PACE intervention
- Control group (Active Comparator): The control group receives usual care, which involves standard CKD education and consultation.
  Interventions: Behavioral: Usual care

INTERVENTIONS:
Behavioral: PACE intervention — "The PACE intervention involves using Line (technological devices) to establish a collaborative group with patients. The researchers will regularly provide reminders to chronic kidney disease patients regarding the importance of nutrition and exercise. They will also provide information on how to adhere to nutritional and exercise regimens, offering praise for consistent performance."
  Arms: PACE intervention
Behavioral: Usual care — Nurses provide routine education and consultation
  Arms: Control group

SUMMARY:
This is a randomized controlled trial study conducted on frail patients with chronic kidney disease(CKD).

DETAILED DESCRIPTION:
The study will be conducted on 120 frail patients with CKD, who will be divided into 2 groups: Group 1, consisting of 60 frail patients, will receive PACE intervention (based on mobile social network support) for 6 months. Group 2, comprising 60 frail patients, will receive usual CKD education and consultation for 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with CKD stage 1 to 5
* Participants with pre-frail and frail conditions.
* Having access to a mobile phone and is capable of using mobile social network application (Line)

Exclusion Criteria:

* Received renal replacement therapy
* Participants achieved TTM stage 5

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2023-10-19 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-09-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- National Cheng Kung University Hospital, Tainan, Taiwan

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients with CKD were recruited from outpatient clinics in hospitals located in southern Taiwan. The eligibility criteria included: (i) age 20 years or older; (ii) diagnosis of CKD stage 1 to 5 for at least 6 months; (iii) identified as frail; (iv) the ability to communicate in Mandarin Chinese or Taiwanese; and (v) willingness to participate in the study. The exclusion criteria were: (i) receiving renal replacement therapy, (ii) a history of mental illness, and (iii) having reached TTM stage 5
Pre-assignment Details: A total of 120 participants were enrolled and assigned to study arms.
Period: Overall Study
Arm/Group | PACE Intervention | Control Group
Started | 60 | 60
Completed | 38 | 58
Not Completed | 22 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PACE Intervention | Control Group | Total
Number analyzed (Participants) | 60 | 60 | 120
Age, Continuous [Mean (Standard Deviation); unit: Years] — Age in years at the time of enrollment, based on medical record documentation.
  Years | 66.70 (13.25) | 69.10 (11.65) | 67.90 (12.48)
Sex: Female, Male [Count of Participants; unit: Participants] — Sex assigned based on patient-reported information at enrollment.
  Participants
    Female | 27 | 30 | 57
    Male | 33 | 30 | 63
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Education Level [Count of Participants; unit: Participants] — Highest education level attained by participant.
  Participants
    Middle school or below | 22 | 30 | 52
    High school or college | 27 | 23 | 50
    University or above | 11 | 7 | 18
Marital Status [Count of Participants; unit: Participants] — Marital status at baseline (e.g., married, single, widowed).
  Participants
    married | 40 | 35 | 75
    single | 10 | 9 | 19
    widowed | 10 | 16 | 26
Living Status [Count of Participants; unit: Participants] — Whether participants lived alone or with others.
  Participants
    lived alone | 11 | 9 | 20
    living with family | 49 | 51 | 100
Estimated Glomerular Filtration Rate (eGFR) [Mean (Standard Deviation); unit: mL/min/1.73m²] — Calculated using MDRD formula.
  mL/min/1.73m² | 36.00 (23.63) | 39.92 (20.34) | 37.96 (22.94)
Serum Albumin [Mean (Standard Deviation); unit: g/dL] — Measured at baseline via blood test. Population: Some participants were excluded from albumin analysis due to missing blood test results at baseline.
  g/dL
    number analyzed (Participants) | 52 | 56 | 108
    (all) | 4.30 (0.53) | 4.28 (0.38) | 4.29 (0.46)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m²] — Calculated as weight (kg) / height (m²). Population: BMI data were missing for one participant in the control group due to incomplete height or weight records at baseline.
  kg/m²
    number analyzed (Participants) | 60 | 59 | 119
    (all) | 25.73 (5.85) | 26.14 (4.74) | 25.93 (5.31)
Hand Grip Strength [Mean (Standard Deviation); unit: kg] — Measured using dynamometer; dominant hand used. Population: Hand grip strength data were missing for three participants due to inability to complete the test or device-related issues at baseline.
  kg
    number analyzed (Participants) | 58 | 59 | 117
    (all) | 23.93 (9.76) | 23.31 (10.82) | 23.62 (10.27)

OUTCOME MEASURES:

1. Primary Outcome: Tilburg Frailty Indicator (TFI)
Description: Frailty was measured using the Tilburg Frailty Indicator (TFI), a 15-item self-reported questionnaire assessing physical, psychological, and social domains. Total score ranges from 0 to 15, with higher scores indicating greater frailty.
Time Frame: Baseline, 3 months, and 6 months post-intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PACE Intervention | Control Group
Number analyzed (Participants) | 60 | 60
score on a scale
  Baseline | 5.38 (2.62) | 4.97 (2.96)
  3 months post-intervention | 4.16 (2.69) | 4.16 (2.37)
  6 months post-intervention | 4.43 (2.81) | 4.74 (2.56)

2. Secondary Outcome: Physical Activity Level Measured by IPAQ-Taiwan
Description: Physical activity was assessed using the International Physical Activity Questionnaire - Taiwan version (IPAQ-Taiwan). Total physical activity score was calculated in MET-minutes/week, including walking, moderate, and vigorous intensity activities.
Time Frame: Baseline, 3 months, and 6 months post-intervention
Measure: Mean (Standard Deviation); unit: MET-minutes/week
Arm/Group | PACE Intervention | Control Group
Number analyzed (Participants) | 60 | 60
MET-minutes/week
  Baseline | 3650.88 (2057.09) | 3971.91 (3647.70)
  3 months post-intervention | 3248.18 (1950.36) | 3891.37 (2747.92)
  6 months post-intervention | 3588.53 (2117.56) | 3259.35 (2140.04)

3. Secondary Outcome: Health-promoting Lifestyle Behaviors (HPLP-II, Taiwan Version)
Description: Lifestyle behaviors were assessed using the HPLP-II, Taiwan version, including six subscales. Scores range from 52 to 208, with higher scores indicating more frequent health-promoting behaviors.
Time Frame: Baseline, 3 months, and 6 months post-intervention
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | PACE Intervention | Control Group
Number analyzed (Participants) | 60 | 60
scores on a scale
  Baseline | 149 (19.93) | 144.6 (21.23)
  3 months post-intervention | 152.93 (19.71) | 149.60 (20.21)
  6 months post-intervention | 149.81 (24.35) | 142.46 (25.72)

4. Secondary Outcome: Nutritional Status Measured by MNA-SF
Description: Nutritional status was assessed using the Mini Nutritional Assessment - Short Form (MNA-SF), a 6-item tool scored 0-14. Higher scores indicate better nutritional status. A score ≥12 is considered normal. The Taiwan version was used.
Time Frame: Baseline, 3 months, and 6 months post-intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PACE Intervention | Control Group
Number analyzed (Participants) | 60 | 60
score on a scale
  Baseline | 12.25 (1.76) | 12.55 (1.60)
  3 months post-intervention | 12.49 (1.30) | 12.59 (1.61)
  6 months post-intervention | 12.42 (1.58) | 12.35 (1.86)

ADVERSE EVENTS:
Time Frame: From baseline to the final follow-up at 6 months post-intervention.
Description: Adverse event data were collected systematically at baseline, 3 months, and 6 months via participant interviews. Definitions aligned with ClinicalTrials.gov.
Arm/Group | PACE Intervention | Control Group
All-Cause Mortality (participants affected / at risk) | 1/60 | 0/60
Serious Adverse Events (participants affected / at risk) | 1/60 | 0/60
Other Adverse Events (participants affected / at risk) | 0/60 | 0/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PACE Intervention (N=60) | Control Group (N=60)
Death, cause unknown (General disorders) | 1 (1) | 0 (0) — The participant was found deceased during the intervention period. No specific cause was determined after clinical evaluation.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PACE Intervention (N=60) | Control Group (N=60)
No other adverse events reported (General disorders) | 0 (0) | 0 (0) — No non-serious adverse events were observed or reported during the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-05-20): https://cdn.clinicaltrials.gov/large-docs/01/NCT06065501/Prot_SAP_000.pdf